CLINICAL TRIAL: NCT04604964
Title: Risk Factors for Anastomotic Leakage in Advanced Ovarian Cancer Surgery: A Large Single Centre Experience
Brief Title: Risk Factors for Anatomic Leakage in Advanced Ovarian Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Other Study IDs: DIPUSVSP-03-02-2032
Record Dates: First submitted 2020-10-11; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Intestinal Anastomotic Leak
Keywords: Recto-sigmoid resection; Advanced Ovarian Cancer; Anastomotic leakage
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing recto-sigmoid resection plus anastomosis: Patients undergoing recto-sigmoid resection and concurrent anastomosis during debulking surgery (primary or interval debunking surgery) for advanced epithelial ovarian cancer.
  Interventions: Other: Evaluation of anastomotic leakage occurrence

INTERVENTIONS:
Other: Evaluation of anastomotic leakage occurrence — Anastomotic leakage was defined as the communication between the intra and extraluminal compartments due to a defect in the integrity of the intestinal wall originating from the staple line of the neo-rectal reservoir between the colon and rectum

SUMMARY:
Cytoreductive surgery is currently the main treatment for advanced epithelial ovarian cancer (AEOC), and the complete disease removal (RT=0) or the achievement of an optimal residual disease (RT < 1 cm) remain the factors with the greatest prognostic impact, both in primary debulking surgery (PDS) and interval debulking surgery (IDS).

To achieve the no residual disease (RT=0), several surgical manoeuvres are often needed both at the upper and lower abdomen, including intestinal resections.

Recto-sigmoid resection is certainly the most frequent of intestinal resections, and it is also the one with the highest risk of complication.

Albeit rare, anastomosis leakage (AL) is a life-threating condition and therefore it is the most feared of intestinal complications.

The aim of this large single-center retrospective study was to assess the AL rate in patients subjected to colorectal resection and anastomosis during primary surgery (PDS or IDS) for advanced ovarian cancer, in a third referral centre for gynecologic oncology with ESGO certification.

In addition, we evaluated several possible pre/intra and post-operative risk factors for AL in order to identify, at an early stage, the population at greatest risk, and attempt to reduce the morbidity and mortality of this severe post-operative complication

DETAILED DESCRIPTION:
The investigators performed a retrospective analysis of the pre-operative, intra-operative and post-operative (surgical outcomes and early complications rate) characteristics, of a series of patients undergoing primary surgery (PDS or IDS) for AEOC at"Fondazione Policlinico Universitario A. Gemelli IRCCS, Università Cattolica del Sacro Cuore, Department of Gynecologic Oncology" between December 2011 and October 2019.

The enrolled population included all patients with histological diagnosis of epithelial ovarian, fallopian or peritoneal cancer (FIGO stage IIB-IVB), judged suitable for surgery by clinicians, and who underwent recto-sigmoid resection and anastomosis with curative intent.

Patients with no evidence of colorectal involvement, and who therefore did not undergo recto-sigmoid resection, or patients with end-colostomy or end-ileostomy were excluded from the study.

Pre-operative clinical variables, surgical features and post-operative outcomes were retrospectively retrieved.

Several system scores, helpful in predicting operative risk, were used to classify patients' physiological status, as the American Society of Anesthesiologists (ASA) score, the Eastern Cooperative Oncology Group-Performance Status (ECOG-PS) and the Age-Adjusted Charlson Comorbidity Index (ACCI).

Patients with an ASA score > 2, ECOG-PS >/= 2 and an ACCI > 2 were considered at high risk of post-operative complications.

Pre-operative albumin level below 30 mg/dl and pre-operative hemoglobin values below 10.0 g/dl were indicative respectively of a severely poor nutritional status and moderate-severe anemia.

Other demographic and surgical variables were recorded: age (< 60 vs >/= 60 year-old), body mass index (BMI) (divided into the following categories: underweight patients: BMI <18, normal weight-overweight: BMI 18-30 and obese patients with BMI >/= 30), International Federation of Gynecology and Obstetrics (FIGO) stage (FIGO stage 2014: </= IIIA vs IIIC-IVB), smoking habit, Ca-125 tumor marker level at initial diagnosis (< 1000 U/mL vs >/= 1000 U/mL), surgical timing (PDS vs IDS), Predictive Index Value (PIV) at initial diagnosis (</= 6 vs > 6), presence of ascites (< 500 mL vs >/= 500 mL), Surgical Complexity Score (SCS) (SCS 1-2 vs SCS 3), estimated blood loss (EBL) (EBL < 500 vs >/= 500 mL) , intra-operative transfusions, additional surgical procedures performed and colorectal resection and anastomosis specific characteristics. The Common Terminology Criteria for Adverse Events v3.0 (CTCAE) was used to classify intra-operative complications (CTCAE 0-1 vs CTCAE >/= 2).

The suspicion of anastomotic leakage (AL), suggested by general clinical signs as abdominal pain or distension, leukocytosis, fever, as well as more specific signs such as emission of gas, pus, or feces via the drains, the laparotomy incision, or the vagina, was ascertained by computed tomography (CT) with rectal contrast enema or simple contrast enema radiography with a water-soluble contrast agent.

The ultimate diagnostic procedure was re-laparotomy with direct verification of AL and/or fecal peritonitis.

Overall survival (OS) was calculated from the date of primary diagnosis to the date of death or to last follow-up visit for the patients still alive.

The primary end-point of the study was to assess the anastomosis leakage rate in patients subjected to colorectal resection and anastomosis during primary surgery (PDS or IDS) for advanced ovarian cancer, in a third referral centre for gynecologic oncology with ESGO certification.

The secondary endpoints were to evaluate the influence of several possible pre/intra and post-operative risk factors on AL in order to identify, at an early stage, the population at greatest risk.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of epithelial ovarian, fallopian or peritoneal cancer
* FIGO stage IIB-IVB
* patients judged suitable for surgery by clinicians
* patients subjected to recto-sigmoid resection and anastomosis with curative intent

Exclusion Criteria:

* Patients with no evidence of colorectal involvement and did not undergo recto-sigmoid resection
* patients with end-colostomy or end-ileostomy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histological diagnosis of epithelial ovarian, fallopian or peritoneal cancer (FIGO stage IIB-IVB), judged suitable for surgery by clinicians, and who underwent recto-sigmoid resection and anastomosis with curative intent between December 2011 and October 2019
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Anastomotic leakage | up to 30 days after surgery
  To assess the anastomotic leakage rate in patients subjected to recto-sigmoid resection during debulking surgery for ovarian cancer

SECONDARY OUTCOMES:
Pre-operative risk factors for anastomotic leakage | just before surgery
  Evaluate the correlation between pre-operative features (age, BMI, ECOG, ACCI, ASA, albumin level, FIGO stage, surgical timing -PDS or IDS, presence of ascites) and the occurrence of anastomotic leakage
Intra-operative risk factors for anastomotic leakage | During surgery
  To evaluate the correlation between surgical procedures (number of bowel resections, hepatic resection, splenectomy, lymphadenectomy, urological procedures as ureteral preimplantation or partial bladder resection, level of inferior mesenteric artery section, distance of the anastomosis from the anal verge, estimated blood loss, intra-operative transfusion, operative time and residual disease) and the occurrence of anastomotic leakage
Post-operative risk factors for anastomotic leakage | up to 30 days after surgery
  To evaluate the correlation between early post-operative complications (post-operative anemia and the occurrence of pancreatic fistula) and the occurrence of anastomotic leakage

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Costantini, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided